CLINICAL TRIAL: NCT01312298
Title: General vs. Intrathecal Anesthesia Fort Total Knee Arthroplasty; a Randomized Clinical Trial
Brief Title: General vs. Intrathecal Anesthesia for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OpHas2011/3; Copenhagen study 2011:1 (Other Grant/Funding Number: Region Skane, SWEDEN)
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-01

CONDITIONS: Arthritis
Keywords: Arthritis; General anaesthesia; Spinal anaesthesia
MeSH Terms: conditions — Arthritis | interventions — Anesthesia, General; Succinylcholine; Air; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Anesthesia (Experimental): Patients allocated to this arm will receive general anesthesia using propofol 10 mg/ml and remifentanil 50 ug/ml in a Target Controlled Infusion (TCI)
  Interventions: Procedure: General anesthesia
- Regional anesthesia (Active Comparator): Patients will receive intrathecal anesthesia
  Interventions: Procedure: Regional anesthesia

INTERVENTIONS:
Procedure: General anesthesia — Patients will receive general anesthesia using propofol 10 mg/ml and remifentanil 50 ug/ml
  Other Names: Suxamethonium 50 mg/ml is used to fascilitate intubation. Ventilation is done using oxygen and air.
  Arms: General Anesthesia
Procedure: Regional anesthesia — Patients will receive intrathecal anesthesia
  Other Names: Patients will receive bupivacaine 5 mg/ml intrathecally. Also the will receive propofol 10 mg/ml to produce a ligth level of sedation.
  Arms: Regional anesthesia

SUMMARY:
Hypothesis: General anesthesia as compared to intrathecal (i.e. spinal anesthesia) anesthesia will result in shorter length of hospital stay for patients undergoing total knee arthroplasty.

Primary endpoint: time from end of surgery until the patient is "street ready"

Secondary endpoints: will general anesthesia produce less postoperative pain as compared to intrathecal anesthesia? Is there any difference in post operative "dizziness" between the groups.

DETAILED DESCRIPTION:
Hypothesis: General anaesthesia compared to intrathecal anaesthesia will give shorter length of hospital stay (LOS) for patients undergoing total knee arthroplasty (TKA).

Primary endpoint: time from end of surgery until the patient meets the discharge criteria.

Secondary endpoints:

1. Will general anesthesia produce less post operative pain?
2. Is there any difference in post operative orthostatic function (dizziness) between the groups?
3. Time until the patient meets the discharge criteria from PACU
4. How many patients will need at least one urinary bladder catheterization?

ELIGIBILITY:
Inclusion Criteria:

1. patients with osteoarthritis scheduled for surgery
2. patients that will require Total Knee Arthroplasty
3. patients over 45 yrs and under 85 yrs
4. patients that understand the given information and are willing to participate in this study
5. patients who have signed the informed consent document

Exclusion Criteria:

1. prior surgery to the same knee
2. patients with a history of stroke or neurological or psychiatric disease that potentially could affect the perception of pain
3. obesity (BMI> 35)
4. active or suspected infection
5. patients taking opioids or steroids
6. patients suffering from rheumatoid arthritis or have a immunological depression.
7. patients who are allergic to any of the drugs being used in this study
8. patients with other severe medical problems that could affect the perioperative course.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
time from end of surgery until patient is "street ready" | within 4 days after surgery
  Time from end of surgery until the patient is street ready will be monitored. If the patient is street ready will be evaluated twice daily each day after the surgery.

SECONDARY OUTCOMES:
Will general anesthesia produce less post operative pain as compared to intrathecal? | 48 hrs after surgery
  Pain will be measured using a visual analogue scale. The patient's own evaluation (questionnaires about quality of life and knee function)
  * Time of post-op department, total time in hospital.
  * Evaluation of patient outcomes, clinical and radiographic evaluation will be done before surgery, after surgery, and after 3 months, after 1year
  * Data collection will be done through normal medical records and patient evaluations collected in a separate file in the clinic. Data is collected and processed by the Research Unit at the orthopedic clinic in Hässleholm.

CONTACTS AND LOCATIONS:
Overall Officials: Sören Toksvig-Larsen, M.D. PhD, Principal Investigator — Dept Ortopedic surgery, Hässleholm Hospital, SWEDEN
Locations (1):
- Dept orthopedic surgery at Hässleholm hospital, Hässlehom, Sweden

REFERENCES:
- [Background] Fowler SJ, Symons J, Sabato S, Myles PS. Epidural analgesia compared with peripheral nerve blockade after major knee surgery: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2008 Feb;100(2):154-64. doi: 10.1093/bja/aem373. PMID 18211990
- [Background] Minto CF, Schnider TW, Shafer SL. Pharmacokinetics and pharmacodynamics of remifentanil. II. Model application. Anesthesiology. 1997 Jan;86(1):24-33. doi: 10.1097/00000542-199701000-00005. PMID 9009936
- [Background] Andersen LO, Husted H, Otte KS, Kristensen BB, Kehlet H. High-volume infiltration analgesia in total knee arthroplasty: a randomized, double-blind, placebo-controlled trial. Acta Anaesthesiol Scand. 2008 Nov;52(10):1331-5. doi: 10.1111/j.1399-6576.2008.01777.x. PMID 19025523